CLINICAL TRIAL: NCT00364052
Title: Prophylactic Therapy for Cytomegalovirus in Liver Transplant Recipients: A Single Center Experience With Oral Ganciclovir Versus Valganciclovir
Brief Title: Prophylactic Therapy for Cytomegalovirus in Liver Transplant Recipients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Oregon Health and Science University (Other)
Other Study IDs: VAL109
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2006-08-17 (Estimated); Status verified 2006-08

CONDITIONS: Liver Transplantation
Keywords: Valganciclovir, Oral Ganciclovir, Liver transplant

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Drug: oral Valganciclovir vs oral Ganciclovir

SUMMARY:
Null Hypothesis:

There is no significant difference in the incidence of CMV infection when using oral valganciclovir or ganciclovir as prophylactic anti-viral therapy.

Alternate Hypothesis:

There exists a significant difference in the incidence of CMV infection when oral valganciclovir is used for CMV prophylaxis rather than oral ganciclovir. A formal hypothesis to be tested should be defined.

DETAILED DESCRIPTION:
The objective for this retrospective clinical study is to describe the incidence of CMV infection in orthoptic liver transplant recipients who receive oral valganciclovir or ganciclovir as their CMV prophylactic anti-viral therapy.

Endpoints:

Primary Endpoint

CMV infection will be characterized as viremia, syndrome or disease by the abovementioned methods for up to one year post-transplantation.

Secondary Endpoints

1. Patient and allograft survival based on donor/recipient CMV status
2. Incidence of graft rejection and loss associated with CMV infection
3. Time to hepatitis C virus (HCV) occurrence
4. Incidence of HSV, EBV and VZV reactivations
5. Severity of HCV occurrence based on biopsy reports based on the Knodell score
6. Safety and tolerability of oral valganciclovir and ganciclovir

ELIGIBILITY:
Inclusion Criteria:

* All liver transplants will be performed at Oregon Health & Science University (OHSU) and the OHSU surgical and medical staff will treat patients.

Exclusion Criteria:

* Portland Veterans Affairs Medical Center liver transplant recipients
* Patients deceased within thirty days of receiving liver allograft
* Patients with low risk of acquiring CMV infection: donor-negative and recipient-negative (D-/R-)
* Patients undergoing re-transplantation
* Lost to follow-up (minimum follow-up is 1 year)
* History of CMV infection or disease
* Anti-CMV therapy within the past 30 d
* Severe, uncontrolled diarrhea or evidence of malabsorption.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2006-08; Study Completion 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Ali J Olyaei, PharmD, Principal Investigator — Oregon Health and Science University